CLINICAL TRIAL: NCT07088744
Title: Comparison of the Sensitivity of Probe-based Confocal Laser Endomicroscopy and Pathological Biopsy Before Endoscopic Submucosal Dissection
Brief Title: Comparison of the Sensitivity of pCLE and Pathological Biopsy Before ESD
Status: Not yet recruiting | Type: Observational
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Zhaoshen Li, Professor, Changhai Hospital
Other Study IDs: Optical biopsy-CLE
Record Dates: First submitted 2025-07-19; First posted 2025-07-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Gastric Cancer (Diagnosis); Gastric High-grade Intraepithelial Neoplasia; Gastric Low-grade Intraepithelial Neoplasia; Gastritis
Keywords: Confocal Laser Endomicroscopy; pathological biopsy
MeSH Terms: conditions — Stomach Neoplasms; Disease; Gastritis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Gastric mucosal biopsy specimens and resected specimens
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

INTERVENTIONS:
Diagnostic Test: Probe-based Confocal Laser Endomicroscopy — Confocal Laser Endomicroscopy (CLE) is an advanced in vivo imaging technique that combines confocal microscopy with endoscopy, enabling real-time, microscopic visualization of tissues at a cellular level during endoscopic procedures. Probe-based CLE (pCLE) can enter the stomach cavity through the biopsy channel of the endoscope and observe the gastric mucosa. All patients scheduled for endoscopic submucosal dissection (ESD) of gastric lesions must undergo probe-based confocal laser endomicroscopy (pCLE) prior to the ESD procedure.
Diagnostic Test: Pathological biopsy — A pathological biopsy is a medical procedure that involves the removal of a small sample of tissue or cells from the body for microscopic examination. It is a crucial diagnostic tool used to identify diseases, particularly cancer, infections, inflammatory conditions, and other abnormalities.

SUMMARY:
Pathological biopsy before endoscopic submucosal dissection (ESD) the gastric lesion plays an important role in differentiating the pathological nature of the lesion and guiding treatment decisions. However, due to the influence of the materials used, the sensitivity of pathological biopsy is not satisfactory. Confocal Laser Endomicroscopy (CLE) is a technology that integrates a confocal microscope into an endoscope. It enables the acquisition of high-resolution microscopic images of the mucosal layer in real-time (with a magnification of up to 1000 times), and it is an optical biopsy technique. It has unique value in the determination of the pathological nature of gastric lesions. The main purpose of this study is to compare the sensitivity of pathological biopsy and CLE in differentiating the pathological nature of gastric lesions.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 18 to 85 years who were scheduled for endoscopic submucosal dissection due to early-stage gastric cancer were consecutively enrolled.

Exclusion Criteria:

* Severe cardiac or pulmonary dysfunction, impaired renal function, coagulopathy, pregnancy or lactation, allergy to fluorescein, and inability to provide informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The absolute indications for curative endoscopic resection (ESD) include moderately and well-differentiated, nonulcerated, mucosal lesions that are ≤2 cm in size. Other relative (expanded) indications for gastric endoscopic submucosal dissection include moderately and well-differentiated superficial cancers that are >2 cm, lesions ≤3 cm with ulceration or that contain early submucosal invasion, and poorly differentiated superficial cancers ≤2 cm in size.
Sampling Method: Non-Probability Sample
Enrollment: 169 (Estimated)
Dates: Start 2025-07-30 (Estimated); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-09-15 (Estimated)

PRIMARY OUTCOMES:
Sensitivity | The pathological results can be obtained within 10 working days after ESD treatment, which can be used for sensitivity calculation.
  Sensitivity, also known as the true positive rate (TPR), refers to the proportion of individuals in the actual patient group that a diagnostic test can correctly identify as positive (i.e., accurately detect cases). High sensitivity means that this detection method can minimize the risk of missed diagnosis to the greatest extent and is suitable for screening diseases (such as infectious diseases and early cancer screening).

SECONDARY OUTCOMES:
Accuracy | The pathological results can be obtained within 10 working days after ESD treatment, which can be used for the calculation of accuracy.
  Accuracy refers to a comprehensive indicator that measures the ability of a medical test or diagnostic method to correctly distinguish between the target disease (such as being ill or not ill). It is the ratio of the sum of true positives and true negatives to the total test population.
Specificity | The pathological results can be obtained within 10 working days after ESD treatment, which can be used for specific calculations.
  Specificity refers to the ability of a diagnostic test to correctly identify individuals who do not have the disease (true negative, TN), that is, the proportion of people who are actually not ill and have a negative test result.

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Guangxi Zhuang Autonomous Region People's Hospital, Nanning, Guangxi
  - Northern Theater Command Hospital, Shenyang, Liaoning
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - The First Affiliated Hospital of Naval Medical University, Shanghai

IPD SHARING:
Plan to Share IPD: No